CLINICAL TRIAL: NCT05140369
Title: Observational Retrospective-Prospective Study on CLL Therapy Approaches in Russia.
Brief Title: CLL Therapy Approaches in Russia
Acronym: CLL registry
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00038
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: This is going to be a non-interventional study (NIS). Assessment of variables will be carried out using data on patient's treatment in real-life clinical setting. Patients should be enrolled into study after evaluation of eligibility criteria by the investigator. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.
  Evaluation of efficacy and safety of any approaches used for CLL/SLL treatment is not the primary objective of this study, though there is no treatment of interest. Study procedures will comply with all the local regulatory requirements regarding AE reporting (pharmacovigilance).
  It is planned to enroll approximately 6000 patients (suggested number of patients on WW~1000 pts, 1L~2750 pts, Relapse/no Response ~2250 pts)

SUMMARY:
This is going to be a non-interventional study (NIS). Assessment of variables will be carried out using data on patient's treatment in real-life clinical setting. Patients should be enrolled into study after evaluation of eligibility criteria by the investigator. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

Evaluation of efficacy and safety of any approaches used for CLL/SLL treatment is not the primary objective of this study, though there is no treatment of interest. Study procedures will comply with all the local regulatory requirements regarding AE reporting (pharmacovigilance).

It is planned to enroll approximately 6000 patients (suggested number of patients on WW~1000 pts, 1L~2750 pts, RR~2250 pts)

During the course of study's prospective part, it is planned to carry out at approximately 5 visits:

(if unscheduled visit performed - the information should be filled on nearest visit).

* Baseline visit: ICF signing, initial patient's data input will be done retrospectively, for patients who are already monitored by investigational site.
* Interim Visits (CRF will be filled every 6 months for therapy receiving patients and every 12 months for WW patients; if a patient transitions from WW to therapy, his/her CRF will be filled every 6 months; all patient's visits should be planned according routine practice and investigator's judgement on individual basis).
* Final visit (data collection on 24 months after enrollment): patient's data input will be done for previously enrolled patients (data update)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability and willing to sign the ICF
* Diagnosed CLL/SLL (including watch and wait stage of disease) according to Russian clinical guides

Exclusion Criteria:

* Patients without CLL/SLL diagnosis
* Age <18 years
* Patients who refused/did not sign the ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected to recruit approximately 6000 patients with CLL/SLL regardless of treatment stage and line.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Sex | Baseline
Date of diagnosis for CLL/SLL | Baseline
Comorbidities | Up to 2 years
ECOG status (0-1/≥2) | Up to 2 years
Rai staging (0-IV) | Up to 2 years
Cytogenetic tests | Up to 2 years
  * TP53 gene mutation status
  * IGHV gene mutation status
  * complex karyotype
  * del13q status

CONTACTS AND LOCATIONS:
Locations (34):
- Russia (34):
  - Research Site, Belgorod
  - Research Site, Bryansk
  - Research Site, Chelyabinsk
  - Research Site, Chita
  - Research Site, Irkutsk
  - Research Site, Kaliningrad
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kirov
  - Research Site, Krasnoyarsk
  - Research Site, Kurgan
  - Research Site, Mahachkala
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Perm
  - Research Site, Petropavlovsk-Kamchatskii
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint-Petesburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Syktyvkar
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Vladimir
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Vologda
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home